CLINICAL TRIAL: NCT03118986
Title: Randomized Controlled Trial of Olanzapine for the Control of Chemotherapy-induced Vomiting in Children Receiving Highly Emetogenic Chemotherapy
Brief Title: RCT of Olanzapine for Control of CIV in Children Receiving Highly Emetogenic Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of California, San Francisco (Other); Children's Mercy Hospital Kansas City (Other); St. Justine's Hospital (Other); Columbia University (Other); Medical University of South Carolina (Other); CancerCare Manitoba (Other); University of North Carolina, Chapel Hill (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Lee Dupuis, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1000053716
Record Dates: First submitted 2017-03-16; First posted 2017-04-18 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-05

CONDITIONS: Vomiting in Infants and/or Children; Nausea; Hematopoietic System--Cancer; Oncology
Keywords: olanzapine; vomiting; children; adolescents; bone marrow transplant; supportive care
MeSH Terms: conditions — Nausea; Neoplasms; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Olanzapine (Active Comparator): Standard antiemetics plus olanzapine
  Interventions: Drug: Olanzapine
- Placebo Oral Tablet (Placebo Comparator): Standard antiemetics plus placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Olanzapine — olanzapine 0.1 mg/kg/dose (maximum 10 mg/dose) by mouth as a single daily dose based on actual body weight
  Arms: Olanzapine
Drug: Placebo Oral Tablet — Placebo tablets that look like olanzapine and will be dosed as if they are olanzapine
  Arms: Placebo Oral Tablet

SUMMARY:
Chemotherapy-induced nausea and vomiting (CINV) are among the most bothersome symptoms during cancer treatment according to children and their parents. Most children receiving highly emetogenic chemotherapy (HEC), including those receiving hematopoietic stem cell transplant (HSCT) conditioning, experience CIV despite receiving antiemetic prophylaxis. Olanzapine improves CINV control in adult cancer patients, has a track record of safe use in children with psychiatric illness, does not interact with chemotherapy and is inexpensive. We hypothesize that the addition of olanzapine to standard antiemetics will improve chemotherapy-induced vomiting (CIV) control in children receiving highly emetogenic chemotherapy

ELIGIBILITY:
Planned receipt of HEC or cyclophosphamide ≥ 1 g/m2/day (≥ 33 mg/kg/day) for cancer treatment or autologous or allogeneic HSCT conditioning.81,82 Examples of HEC are: busulfan IV (myeloablative dosing), carboplatin ≥175mg/m²/dose, cisplatin ≥12mg/m²/dose, cytarabine ≥3g/m²/day, melphalan >140mg/m², methotrexate ≥12g/m²/dose and thiotepa ≥300mg/m²/dose.

Plan for inpatient admission from administration of first study drug dose until 24 hours following administration of last study drug dose.

Body weight of at least 12.5 kg

2.5 to < 18 years of age. Note that the minimum age requirement corresponds to an approximate body weight of 12.5 kg.

Samples for all laboratory tests will be obtained within one week prior to administration of the first chemotherapy dose of the study chemotherapy block or the first HSCT conditioning dose:

* Plasma creatinine within 1.5 times the upper limit of normal for age.
* Amylase within age-appropriate limits
* Plasma conjugated bilirubin within ≤ 3x upper limit of normal for age unless attributable to Gilbert's Syndrome
* ALT ≤ 5x upper limit of normal for age

Baseline ECG within the month prior to study drug administration without known clinically significant abnormalities including pathologic prolongation of QTc

A plan for scheduled, round-the-clock receipt of ondansetron, granisetron or palonosetron for antiemetic prophylaxis during administration of chemotherapy or HSCT conditioning.

Negative pregnancy test if female of childbearing potential

Patients of childbearing potential must consent to use adequate contraception (males and females) or agree to practice abstinence

Parent or child able to speak a language in which the (modified Pediatric Adverse Event Rating Scale (PAERS) is available.

Optional: Child participants in the optional assessment of nausea severity must be 4 to 18 years of age. Child and a parent/guardian must be English, Spanish or French-speaking. The Pediatric Nausea Assessment Tool58 (PeNAT) is validated in English-speaking children 4 to 18 years old with an English-speaking parent/guardian and has been translated into Spanish and French. The MAT is available in English, Spanish and French.

Ages: 30 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Rate of CIV control during the acute phase | up to 8 days
  Complete CIV control is no vomiting/retching and no use of breakthrough antiemetic agents during phase
Rate of CIV control during the acute phase | up to 8 days
  Partial control is defined as no more than two vomits or retches during any 24-hr period

SECONDARY OUTCOMES:
complete and partial CINV control | up to 1 month
  Complete CIV control is no vomiting/retching and no use of breakthrough antiemetic agents during phase, Partial control is defined as no more than two vomits or retches during any 24-hr period
Safety profile of olanzapine based on toxicities | up to 1 month
  Based on descriptive statistics on reported toxicities.
Safety profile of olanzapine based on weight | up to 1 month
  Based on descriptive statistics on reported body weight
Safety profile of olanzapine based on Pediatric Adverse Event Rating Scale (PAERs) | up to 1 month
  Based on descriptive statistics on reported PAERs, will describe the most reported and most bothersome adverse events reported in the PAERs questionnaire.
Safety profile of olanzapine based on prolactin | up to 1 month
  Based on descriptive statistics on reported prolactin, will report incidence of abnormal prolactin values comparing the two arms
Safety profile of olanzapine based on amylase | up to 1 month
  Based on descriptive statistics on reported amylase, will report incidence of abnormal amylase values comparing the two arms
Safety profile of olanzapine based on creatine phophotase | up to 1 month
  Based on descriptive statistics on reported creatine phophotase, will report incidence of abnormal creatine phophotase values comparing the two arms
Safety profile of olanzapine based on triglycerides | up to 1 month
  Based on descriptive statistics on reported triglycerides, will report incidence of abnormal triglyceride values comparing the two arms
Impact of olanzapine on HSCT outcomes on incidence of veno-occlusive disease | From first HSCT conditioning dose until 100 days post-HSCT
  Looking at incidence of veno-occlusive disease
Impact of olanzapine on HSCT outcomes on incidence of GVHD | From first HSCT conditioning dose until 100 days post-HSCT
  Looking at incidence of GVHD between the two arms
Impact of olanzapine on HSCT outcomes on severity of GVHD | From first HSCT conditioning dose until 100 days post-HSCT
  Comparing the incidence of the different maximal grades of GVHD between the two arms
Association between PeNAT and MASCC Antiemesis Tool (MAT) scores | up to 1 month
  taking maximum daily PeNAT scale score and maximum nausea experience in MAT will estimate the degree of association between PeNAT and MAT

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dupuis, RPh, PhD, Principal Investigator — The Hospital for Sick Children; Muhammad Ali, MD, Principal Investigator — The Hospital for Sick Children
Locations (10):
- United States (6):
  - University of California, San Francisco, California
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University/Morgan Stanley Children's Hospital, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
- Canada (3):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine,, Montreal, Quebec
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dupuis LL, Taddio A, Kerr EN, Kelly A, MacKeigan L. Development and validation of the pediatric nausea assessment tool for use in children receiving antineoplastic agents. Pharmacotherapy. 2006 Sep;26(9):1221-31. doi: 10.1592/phco.26.9.1221. PMID 16945043